CLINICAL TRIAL: NCT02604095
Title: Effect of Melatonin on Body Composition, Glucose Metabolism and Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Professor, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Melatonin
Record Dates: First submitted 2015-11-05; First posted 2015-11-13 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Acanthosis Nigricans; Obesity
Keywords: Acanthosis nigricans; Obesity
MeSH Terms: conditions — Acanthosis Nigricans; Obesity | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melatonin (Experimental): Take one table at bedtime.
  Interventions: Dietary Supplement: melatonin

INTERVENTIONS:
Dietary Supplement: melatonin — Take one tablet (containing melatonin 3mg, calcium 52mg, vitamin B6 5mg) at bedtime everyday for 12 weeks.

SUMMARY:
Effect of Melatonin on Body Composition, Glucose Metabolism and Lipid Metabolism.

DETAILED DESCRIPTION:
The effect of Melatonin on Body Composition, Glucose Metabolism and Lipid Metabolism in patient with obesity and acanthuses nigrican.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-60 years old;
* BMI ≥ 28 kg/m2；
* With acanthosis nigricans。

Exclusion Criteria:

* With liver, kidney, gastrointestinal or other major organic serious diseases, cancer, lactating women, pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
insulin resistance index | 12 weeks
  HOMA-IR:serum fasting insulin(mmol/L) × serum fasting glucose(mmol/L)/22.5

SECONDARY OUTCOMES:
Blood pressure | 12 weeks
  Systolic blood pressure (mmHg) and diastolic blood pressure (mmHg)
Body weight | 12 weeks
  Body weight (kg)
Body fat | 12 weeks
  Body fat (%)
Neck circumference | 12 weeks
  Neck circumference (cm)
Waist circumference | 12 weeks
  Waist circumference (cm)
Total Cholesterol | 12 weeks
  Total Cholesterol (mmol/L)
Triglyceride | 12 weeks
  Triglyceride (mmol/L)
Low Density Lipoprotein | 12 weeks
  Low Density Lipoprotein (mmol/L)
High Density Lipoprotein | 12 weeks
  High Density Lipoprotein (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Ph.D, Study Director — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People' Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Sun H, Wang X, Chen J, Gusdon AM, Song K, Li L, Qu S. Melatonin Treatment Improves Insulin Resistance and Pigmentation in Obese Patients with Acanthosis Nigricans. Int J Endocrinol. 2018 Mar 12;2018:2304746. doi: 10.1155/2018/2304746. eCollection 2018. PMID 29706998